CLINICAL TRIAL: NCT06576375
Title: Efficacy of Dapagliflozin Versus Metformin in Polycystic Ovary Syndrome: A Prospective Comparative Randomized Blinded Trial.
Brief Title: Efficacy of Dapagliflozin Versus Metformin in Polycystic Ovary Syndrome
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Future University in Egypt (Other)
Collaborators: October 6 University (Other)
Responsible Party: Principal Investigator, Nouran Omar El Said, Lecturer in Pharmacy Practice & Clinical Pharmacy, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRC-Ph-2307003
Record Dates: First submitted 2024-08-23; First posted 2024-08-28 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-08

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — dapagliflozin; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin (Active Comparator): Patients will receive Dapagliflozin 10 mg once daily orally for 12 weeks (Forxiga® AstraZeneca company)
  Interventions: Drug: Dapagliflozin
- Metformin (Active Comparator): Patients will receive Metformin 1000 mg once daily orally for 12 weeks (control group) (Glucophage® Merck company)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Dapagliflozin — oral Dapagliflozin
  Arms: Dapagliflozin
Drug: Metformin — oral metformin
  Arms: Metformin

SUMMARY:
In PCOS (Polycystic Ovary Syndrome), studies have found impaired incretin secretion and activity, particularly in overweight/obese individuals.

Conflicting results exist regarding glucagon-like peptide-1(GLP-1) levels in PCOS patients, with studies reporting reduced, normal, or increased levels. Incretin-based therapy has been suggested as a potential treatment to reverse prediabetes risk by preserving β-cell function in patients with impaired fasting glucose(IFG and impaired glucose tolerance(IGT). The study aims to compare the efficacy of Dapagliflozin to Metformin for the treatment of non-diabetic patients with polycystic ovary syndrome (PCOS).

DETAILED DESCRIPTION:
Incretins such as glucagon-like peptide-1(GLP-1) are gut hormones secreted after meals that enhance insulin secretion and help maintain glucose homeostasis.They also reduce hepatic glucagon release, slow gastric emptying, and suppress appetite, aiding in weight control and glycemic management.In PCOS (Polycystic Ovary Syndrome), studies have found impaired incretin secretion and activity, particularly in overweight/obese individuals.Conflicting results exist regarding GLP-1 levels in PCOS patients, with studies reporting reduced, normal, or increased levels.After an oral glucose tolerance test, increased GIP and lower GLP-1 concentrations have been observed in women with PCOS.

Reduced GLP-1 levels are also associated with impaired glucose tolerance (IGT) and impaired fasting glucose (IFG), which are early indicators of prediabetes and potential progression to Type 2 Diabetes Mellitus.Incretin-based therapy has been suggested as a potential treatment to reverse prediabetes risk by preserving β-cell function in patients with IFG and IGT. The study aims to compare the efficacy of Dapagliflozin to Metformin for treatment of non-diabetic patients with polycystic ovary syndrome (PCOS).

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with PCOS according to Rotterdam 2003 criteria National Institute of Health criteria.
* Age: >18 <40 years.
* Infertile women (primary or secondary infertility)

Exclusion Criteria:

* Patients with history of diabetes mellitus (Type 1 or 2).
* Patients with liver or renal dysfunction; inflammatory diseases; autoimmune disease; cancer, acute cardiovascular event within last three months and uncontrolled endocrine or metabolic disease.
* Use of hormonal medications, lipid-lowering (statins, etc.), anti-obesity drugs or weight loss medications (prescription or OTC) and medications known to exacerbate glucose tolerance (such as isotretinoin, hormonal contraceptives, glucocorticoids, anabolic steroids) stopped for at least 8 weeks. Use of anti-androgens that act peripherally to reduce hirsutism such as 5-alpha reductase inhibitors stopped for at least 4 weeks.
* Patients at risk for volume depletion due to co-existing conditions or concomitant medications, such as loop diuretics should have careful monitoring of their volume status.
* Presence of hypersensitivity to dapagliflozin or other Sodium/glucose cotransporter 2 (SGLT2) inhibitors (e.g. anaphylaxis, angioedema, exfoliative skin conditions).
* Use of Metformin, Thiazolidinediones, glucagon-like peptide-1 (GLP-1) receptor agonists, DPP-4 inhibitors, SGLT2 inhibitors
* Eating disorders (anorexia, bulimia) or gastrointestinal disorders.
* Having a history of bariatric surgery.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Fertility parameters- Luteinizing hormone | 3-6 months
  Luteinizing hormone (LH) in IU/L
Fertility parameters-Follicle-stimulating hormone | 3-6 months
  Follicle-stimulating hormone (FSH) in mIU/mL
Fertility parameters-Free androgen index | 3-6 months
  Free androgen index [ Time Frame: 3-6 months]
Fertility parameters-Total testosterone | 3-6 months
  Total testosterone in ng/dL
Transvaginal ultrasonography | 3-6 months
  disappearance of PCOS
Menstrual diaries | 3-6 months
  Menstruation pattern

SECONDARY OUTCOMES:
Metabolic parameters | 3-6 months
  Fasting blood glucose (FBG) in mg/dL

CONTACTS AND LOCATIONS:
Locations (1):
- October 6 University Hospital, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No